CLINICAL TRIAL: NCT05741554
Title: LOw Grade Serous Ovarian Carcinoma and Uterine Involvement : Should hYSTerectomy be the Rule
Acronym: LOGYST
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 22-5035; 69HCL23_0175 (Other: HCL)
Record Dates: First submitted 2023-02-14; First posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Serous Ovarian Carcinoma; Low Grade Serous Ovarian Carcinoma
Keywords: Serous ovarian carcinoma; Low grade serous ovarian carcinoma; Fertility sparring surgery; Hysterectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Myometrial involvement: Myometrial involvement by cancer metastasis after pathology examination
  Interventions: Other: Rate of myometrial involvement in the population of 28 low grade serous ovarian carcinoma.
- No myometrial involvement: Absence of myometrial involvement by cancer metastasis after pathology examination
  Interventions: Other: Rate of myometrial involvement in the population of 28 low grade serous ovarian carcinoma.

INTERVENTIONS:
Other: Rate of myometrial involvement in the population of 28 low grade serous ovarian carcinoma. — Presence of uterine myometrial metastasis at pathology examination after cytoreductive surgery

SUMMARY:
Investigators studied a population of 28 low grade serous ovarian carcinoma treated in Hospices civils de Lyon between 2000 and 2022. The primary objective is to determinate the rate of myometrial involvement by the cancer at pathology examination. Then, investigators compared patients with or without myometrial involvement : survival parameters, predictive factors of myometrial involvement (age, CA 125 level, surgery characteristics, pathology characteristics).

ELIGIBILITY:
* Inclusion Criteria :

  * 18 years old or more
  * low grade serous ovarian cancer (MDACC classification)
  * Grade 1 serous ovarian carcinoma (Silverberg classification)
* Exclusion Criteria :

  * no sufficient data available
  * grade 2 and 3 serous ovarian carcinoma

Sex: Female
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: All patients treated in hospices Civils de Lyon for a Low grade serous ovarian cancer between January 2000 and May 2022
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Percentage of myometrial involvement | After pathology examination, average 2 to 3 weeks after cytoreductive surgery
  Myometrial involvement after pathology examination

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices civils de Lyon, Lyon, France